CLINICAL TRIAL: NCT04582214
Title: A Pilot Study of the Use of Oscillation and Lung Expansion (OLE) Therapy in Patients Hospitalized With COVID-19
Brief Title: Oscillation and Lung Expansion Therapy in Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hill-Rom (Industry)
Collaborators: Emory University (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-RR-2020-002
Record Dates: First submitted 2020-10-06; First posted 2020-10-09 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Oscillation and Lung Expansion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The active treatment group will consist of patients who are treated OLE therapy while on heated high-flow oxygen therapy. Results from subjects in the active treatment group will be compared to retrospectively collected results from patients treated with standard care with no OLE therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OLE Therapy with The MetaNeb® System (Experimental): Subjects in the active treatment group will receive OLE therapy with The MetaNeb® System following the labeled instructions for the device.
  Interventions: Device: MetaNeb® System
- Control Group (No Intervention): The airway clearance regimen for subjects in the control group will be collected from the medical record.This information will be retrospectively collected from patients treated with standard care with no OLE therapy. Subjects in the control group will be identified from the population of patients previously admitted to the two study sites with COVID-19 infection who required invasive mechanical ventilation but were not treated with OLE therapy.

INTERVENTIONS:
Device: MetaNeb® System — The intervention device use in this study is The MetaNeb® System (Hill-Rom; St. Paul, MN). It is an FDA 510k cleared device (k124032), powered by compressed gas, that delivers oscillation and lung expansion (OLE) therapy using both continuous high-frequency oscillation (CHFO) and continuous positive expiratory pressure (CPEP). The device also provides supplemental oxygen when used with compressed oxygen and can deliver aerosol therapy during CPEP and/or CHFO. The therapy is indicated for mobilization of secretions, lung expansion therapy and the treatment and prevention of pulmonary atelectasis. The device also provides supplemental oxygen when used with compressed oxygen.
  Arms: OLE Therapy with The MetaNeb® System

SUMMARY:
A Pilot Study of the Use of Oscillation and Lung Expansion (OLE) Therapy in Patients Hospitalized with COVID-19

DETAILED DESCRIPTION:
This is a randomized prospective open-label cohort study in patients with COVID-19 to evaluate the impact of Oscillation and Lung Expansion (OLE) therapy using The MetaNeb® System on the hospital length of stay in patients hospitalized and receiving heated high-flow oxygen therapy for COVID-19 infection. The active treatment group will consist of patients who are treated OLE therapy while on heated high-flow oxygen therapy .

Results from subjects in the active treatment group will be compared to results from patients treated with standard care with no OLE therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years of age)
* Tested positive or person under investigation (PUI) for COVID-19 infection
* Currently require heated high-flow oxygen therapy to maintain SaO2 > 90 %
* Signed informed consent (phone consent)
* Heated high-flow oxygen initiated within the past 72 hours

Exclusion Criteria:

* Serious medical condition that, in the investigator's judgment, precludes the patient's safe participation in the study
* Pressure related risk for pneumothorax
* Patient inability or unwillingness to tolerate OLE therapy
* Staff unavailable or unable to deliver therapy
* Current requirement for mechanical ventilation or expected requirement for mechanical ventilation within the next 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Length of Stay | Time frame begins when the patient is first started on heated high-flow oxygen therapy and ends when they are ready for discharge from the hospital. Expected time is a a few days but not expected to exceed 3 weeks.
  Number of days/hours the patient is in the hospital after initiation of high-flow oxygen therapy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No